CLINICAL TRIAL: NCT03095287
Title: A Multicenter Phase 2 Open-Label, Single-Arm, Prospective, Interventional Study of Plasma-Derived Factor VIII/VWF (Alphanate®) in Immune Tolerance Induction Therapy in Subjects With Congenital Hemophilia A
Brief Title: Alphanate in Immune Tolerance Induction Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to limited enrollment (non-safety related decision)
Sponsor: Grifols Therapeutics LLC (Industry)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBI1406; 2015-005524-26 (EudraCT Number)
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Hemophilia A, Congenital
Keywords: Factor VIII; von Willebrand Factor; Plasma-derived; Inhibitors; Immune tolerance induction (ITI); Antibodies; Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII, von Willebrand factor drug combination; von Willebrand Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alphanate (Experimental): Participants were to receive alphanate 100 International Units (IU/kg/day) for up to 33 months in Immune tolerance induction (ITI) Treatment Phase. The dose could be increased up to 200 IU/kg/day based on Investigator's discretion. Following ITI Treatment Phase, participants were to enter the Prophylactic Phase where alphanate dose was to be tapered down in a step wise manner to reach a final prophylactic dose of 50 IU/kg every other day or 3 times per week, at the investigator's discretion.
  Interventions: Biological: Alphanate

INTERVENTIONS:
Biological: Alphanate — Bolus IV injection.
  Other Names: Factor VIII/von Willebrand Factor

SUMMARY:
This is a multicenter, multinational, prospective, single-arm, nonrandomized, open-label study, planned in of approximately 25 male participants with congenital hemophilia A who will receive their first (primary) immune tolerance induction (ITI) treatment with alphanate.

The study consists of 2 phases:

* An ITI Treatment Phase in which all eligible participants will receive ITI treatment with alphanate for a period of up to 33 months. Upon confirmation of complete immune tolerization, participants will then enter a 12-month Prophylactic Phase. If, after 33 months of ITI, a participants has achieved partial immune tolerance, the participants will enter a 12-month Prophylactic Phase.
* A 12-month Prophylactic Phase for all participants who meet the criteria for complete or partial success to continue on a prophylactic dosing regimen of alphanate. Due to limited enrollment, this study was early terminated.

DETAILED DESCRIPTION:
Male participants <12 years of age with an inhibitor titer >0.6 to <10 Bethesda Units (BU) will be screened before the planned start of ITI treatment. Participants continuing to meet the entrance criteria will enter the ITI Treatment Phase and receive daily doses of alphanate 100 IU/kg/day for up to 33 months, with a one-time option to increase to a dosing regimen of 200 IU/kg/day at any time after 90 days of ITI treatment.

Participants will continue to receive their daily alphanate dose for up to 33 months until the titer is negative (<0.6 BU) on 2 consecutive assessments and treatment success is confirmed by FVIII:C pharmacokinetic assessments, at which time they will enter the 12-month Prophylactic Phase.

In addition, participants who have achieved partial immune tolerance at the completion of 33 months of ITI treatment will enter the 12-month Prophylactic Phase. Participants who do not achieve partial immune tolerance at the completion of 33 months of ITI treatment will be discontinued as treatment failures.

The Prophylactic Phase begins with an 8-week taper period for participants tolerized with 100 IU/kg/day or with a 12-week taper period for participants tolerized with 200 IU/kg/day to bring the dose down in a step-wise manner to a prophylactic dose of alphanate 50 IU/kg every other day or 3 times per week, at the investigator's discretion. During the Prophylactic Phase, participants will be monitored monthly for the first 4 months and then every 2 months for the remaining 8 months to assess sustainability of immune tolerance. Due to limited enrollment, this study was early terminated.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a documented diagnosis of severe congenital hemophilia A with FVIII:C <1% of normal.
* The subject is a male <12 years (and at least 2 years of age if in India) at the Baseline Visit.
* The subject's documented historical peak inhibitor titer is ≥5 BU and ≤200 BU.
* The subject has an inhibitor titer >0.6 BU and <10 BU at Screening.
* The subject has had a delay ≤24 months from the date of diagnosis of the inhibitor to the start of the subject's ITI treatment.

Exclusion Criteria:

* The subject has acquired factor VIII (FVIII) deficiency.
* The subject has previously received ITI treatment.
* The subject has a recent (within 1 month) history of central line infection at the time of Screening.
* The subject has a high risk of cardiovascular, cerebrovascular, or thromboembolic event as judged by the investigator.
* The subject is currently undergoing treatment with immunosuppressive drugs (eg, systemic corticosteroids), azathioprine, cyclophosphamide, high dose immunoglobulin, interferon, or the use of a protein A column or plasmapheresis and is unwilling to discontinue these treatments starting at the screening visit.
* The subject has a known infection with human immunodeficiency virus (HIV) or has clinical signs and symptoms consistent with current HIV infection.
* The subject has a known previous infection with hepatitis B virus (HBV) or hepatitis C virus (HCV) or has clinical signs and symptoms consistent with current HBV or HCV infection.
* The subject has significant proteinuria, has a history of acute renal failure or severe renal impairment (blood urea nitrogen or creatinine >2 times the upper limit of normal), or is receiving dialysis at Screening.
* The subject has a value of aspartate transaminase or alanine aminotransferase >2 times the upper limit of normal at Screening.
* The subject has clinical evidence of any significant acute or chronic disease that, in the opinion of the investigator, may interfere with successful completion of the trial or place the subject at undue medical risk.
* The subject has a history of anaphylaxis or severe systemic reaction to any plasma derived or other blood products.

Max Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (8):
  - Emory University, Atlanta, Georgia
  - University of Kentucky, Lexington, Kentucky
  - Childrens Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Robert Wood Johnson Medical Group, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center & Children's Hospital of New Jersey, Newark, New Jersey
  - University of North Carolina at Chapel Hill, Hemophilia and Thrombosis Center, Chapel Hill, North Carolina
  - Seattle Children's Hospital, Seattle Children's Research Institute, Seattle, Washington
- McMaster Children's Hospital, Hamilton, Ontario, Canada
- India (2):
  - Lokmanya Tilak Municipal Medical College & General Hospital, Mumbai, Maharashtra
  - B. J. Govt. Medical College & Sassoon Hospital, Pune
- Italy (3):
  - A.O.U. Santa Maria della Misericordia Perugia, Perugia, Umbria
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Universita degli Studi di Roma La Sapienza, Roma
- Russia (3):
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - FGUs Hospital - Kirov Scientific Research Institute, Kirov
  - Center for Hemophilia Treatment St.-Petersburg, Saint Petersburg
- Spain (3):
  - Hospital Universitari i Politecnic La Fe, Valencia, Autonomous Community of Valencia
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at two sites in India from 03 January 2018 (first participant enrolled to receive the study drug) to 18 September 2020 (last participant completed).
Pre-assignment Details: Male participants with diagnosis of Congenital Hemophilia A were enrolled in a single arm to receive alphanate. The study was to be conducted in 2 phases: Immune Tolerance Induction Phase followed by Prophylactic Phase. However, due to the limited enrollment, the study was terminated prior to the start of Prophylactic Phase.
Groups:
- Alphanate: Participants entered the immune tolerance induction (ITI) phase and received alphanate IV at a starting dose of 100 IU/kg/day. Dose could be uptitrated to 200 IU/kg/day based on investigator's discretion. The maximum duration of treatment was 32 months and 2 weeks.
Period: Overall Study
Arm/Group | Alphanate
Started | 2
Completed | 0
Not Completed | 2
Not completed — Treatment Failure | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | Alphanate
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Complete Immune Tolerance Within 33 Months of Initiation of Immune Tolerance Induction (ITI) Treatment Phase
Description: Complete immune tolerance was defined as the participants achieving 2 consecutive undetectable inhibitor titers (<0.6 BU) performed within 2 weeks of each other, Factor VIII activity (FVIII:C) in vivo plasma recovery ≥66% of the predicted normal value and FVIII:C half-life ≥6 hours after a 72-hour FVIII treatment-free period.
Time Frame: Up to 32.5 months
Population: Data for this outcome measure was not collected and analysed, as the study was early terminated by the sponsor due to limited enrollment (non-safety related decision).
Arm/Group | Alphanate
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage of Participants Who Achieved Either Complete or Partial Immune Tolerance Within 33 Months of Initiation of ITI Treatment Phase
Description: Complete immune tolerance was defined as the participants achieving 2 consecutive undetectable inhibitor titers (<0.6 BU) performed within 2 weeks of each other, Factor VIII activity (FVIII:C) in vivo plasma recovery ≥66% of the predicted normal value and FVIII:C half-life ≥6 hours after a 72-hour FVIII treatment-free period. Partial immune tolerance was defined as participants achieving reduction of inhibitor titer to <5 BU confirmed at 2 consecutive assessments within 2 weeks of each other, FVIII:C in vivo plasma recovery of <66% of the predicted normal value or FVIII:C half-life of <6 hours after a 72-hour FVIII treatment-free period and clinical response to FVIII therapy.
Time Frame: Up to 32.5 months
Population: as for outcome 1
Arm/Group | Alphanate
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants Who Achieved Complete or Partial Immune Tolerance Without Relapse During the Prophylactic Phase
Description: Relapse during the prophylactic phase for participants who have achieved complete immune tolerance was defined as a return of FVIII inhibitor titer to detectable levels (≥0.6 BU) or FVIII:C recovery <66% of the predicted normal value or FVIII:C half-life <6 hours, confirmed by repeat assessment within approximately 2 weeks. Relapse for participants who have achieved partial immune tolerance was defined as an increase of FVIII inhibitor titer to ≥5 BU, confirmed by repeat assessment within approximately 2 weeks.
Time Frame: 12 months during prophylactic phase
Population: as for outcome 1
Arm/Group | Alphanate
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Bleeding Events During ITI Treatment Phase and Prophylactic Phase
Description: Annualized frequencies of bleeding events during the ITI Treatment Phase and the Prophylactic Phase
Time Frame: Up to 32.5 months
Population: This study was terminated, and the data is not reported for this outcome measure to maintain participant's confidentiality.
Arm/Group | Alphanate
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Treatment-emergent Adverse Events
Description: Incidence of treatment-emergent adverse events during the ITI Treatment Phase and Prophylactic Phase
Time Frame: Up to 32.5 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From first dose up to 32.5 months
Description: Safety population included all participants who received any amount of alphanate.
Groups:
- Alphanate: Participants entered the ITI phase and received alphanate IV at a starting dose of 100 IU/kg/day. Dose could be uptitrated to 200 IU/kg/day based on investigator's discretion. The maximum duration of treatment was 32 months and 2 weeks.
Arm/Group | Alphanate
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alphanate (N=2)
Lower respiratory tract infection (Infections and infestations) | 1
Subdural hemorrhage (Injury, poisoning and procedural complications) | 1
Device related infection (Infections and infestations) | 1
Hepatitis C Antibody positive (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alphanate (N=2)
Thrombophlebitis (Vascular disorders) | 1
Pyrexia (General disorders) | 2
Transaminases increased (Investigations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Headache (Nervous system disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Varicella (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Nasopharyngitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT03095287/Prot_SAP_001.pdf